CLINICAL TRIAL: NCT02099617
Title: Efficacy and Safety of New Generation Drug Eluting Stents Associated With an Ultra Short Duration of Dual Antiplatelet Therapy. Design of the Short Duration of Dual antiplatElet Therapy With SyNergy II Stent in Patients Older Than 75 Years Undergoing Percutaneous Coronary Revascularization.
Acronym: SENIOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ceric Sàrl (Industry)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-389
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2024-01-16 (Actual); Status verified 2017-05

CONDITIONS: Stable Angina; Silent Myocardial Ischemia; Acute Coronary Syndrome
MeSH Terms: conditions — Angina, Stable; Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Eluting Stent (Experimental): Synergy II
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Synergy II stent
- Bare Metal Stent (Active Comparator): Omega or Rebel
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Omega stent; Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Rebel stent

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Synergy II stent
  Arms: Drug Eluting Stent
Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Omega stent
  Arms: Bare Metal Stent
Procedure: Percutaneous Coronary Intervention (PCI) with short DAPT duration with Rebel stent
  Arms: Bare Metal Stent

SUMMARY:
The main objective of the SENIOR study is to establish the efficacy and safety of the everolimus eluting stent with a biodegradable abluminal polymer (SYNERGY II) associated with a short dual antiplatelet therapy (DAPT) in patients ≥75 years old, suffering from stable angina, silent ischemia (1 month DAPT) or acute coronary syndromes (6 months DAPT) related to significant coronary artery disease and requiring percutaneous coronary intervention. The primary end point is to demonstrate that SYNERGY II in patients ≥75 years old is associated with a lower rate of the composite rate of major cardiovascular and cerebrovascular events (all-cause death, myocardial infarction, stroke, ischemia-driven target lesion revascularization) and a similar risk of stent thrombosis than bare metal stent at one year.

ELIGIBILITY:
Inclusion Criteria:

* 1- Patient is ≥ 75 years old
* 2- One or more significant coronary artery stenosis is/are present (defined as ≥70% by visual assessment or ≥50% with Fractional Flow Reserve <0.80) or a left main coronary stenosis ≥50% by visual assessment) suitable for PCI with one of the following present:
* a -Silent ischemia,
* stress-induced myocardial ischemia ≥ 10% of myocardium in a asymptomatic patient or
* stress-induced myocardial ischemia < 10% of myocardium AND FFR (Fractional Flow Reserve) ≤0.80 or
* b - Stable angina, in a patient with objective ischemia despite optimal medical therapy or
* c - acute coronary syndrome including: unstable angina, non ST- and ST elevation myocardial infarction.
* 3- All patients must also sign informed consent as per local law and comply with all study process during follow up for at least one year.

Exclusion Criteria:

* 1- The subject is not eligible for randomization if ANY of the following is present:
* 2- Indication for myocardial revascularization by coronary artery bypass grafting,
* 3- Subjects unable to tolerate, obtain or comply with dual antiplatelet therapy for at least one month (stable angina or silent ischemia) or at least six month (acute coronary syndrome),
* 4- Subjects requiring additional surgery (cardiac or non-cardiac) within one month,
* 5- Non cardiac co-morbidities with life expectancy less than 1 year,
* 6- Prior hemorrhagic stroke,
* 7- Known allergy to aspirin or P2Y12 inhibitors,
* 8- At least one contra indication to ALL the authorized P2Y12 inhibitors at the requested dose (in case of contra indication to only one of two of the P2Y12 inhibitors, the investigators are allowed to use the P2Y12 inhibitors for which no allergy is known).
* 9- Silent ischemia <10% of the myocardium with FFR ≥0.80.
* 10- Participation in another clinical trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Composite measure of MACCEs (Major Adverse Cardiac and Cerebrovascular Events) | 12 months
  all-cause death, non fatal myocardial infarction, non fatal stroke, ischemia-driven target lesion revascularization.

SECONDARY OUTCOMES:
Primary endpoint | 30 days, 180 days, 2 years
All revascularizations | 30 days, 180 days, 1 year, 2 years
  All target lesion revascularization, all target vessel revascularization, all non target vessel revascularization
Complete revascularization | Baseline procedure
  anatomic and functional
Net benefit | 30 days, 180 daysn 1 year, 2 years
  association of composite events (all cause mortality, myocardial infarction, stroke, ischemia driven target lesion revascularization, and major bleedings)
Major bleedings complications | 30 days, 180 days, 1 year, 2 years
  type 2, 3 and 5 BARC definition)
Stent thombosis | 30 days, 1 year, 2 years
  according to the definition of ARC symptomatic or asymptomatic (definite + probable)
QoL | 12 months, 24 months
Depression scale | 12 months, 24 months
Cost effectiveness | 12 months

CONTACTS AND LOCATIONS:
Locations (44):
- Belgium (4):
  - CHU St Pierre, Brussels
  - Centre Hospitalier de Jolimont, La Louvière
  - UZ Leuven, Leuven
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
- Finland (2):
  - Oulu University Hospital, Oulu
  - Heary Center - Satakunta Centyral Hospital, Pori
- France (11):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Henri Mondor, Créteil
  - Hôpital de la Timone, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - Polyclinique les Fleurs, Ollioules
  - Hôpital Lariboisière, Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Privé Claude Galien, Quincy-sous-Sénart
  - CHU Toulouse Rangueil, Toulouse
- ARNAS civico, Palermo, Italy
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- University Clinic of Cardiology - Medical Faculty, Skopje, North Macedonia
- Spain (13):
  - Hospital universitario Marquès de Valdecilla, Santander, Cantabria
  - Hospital San Juan de Alicante, Alicante, Valencia
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universati Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de la Santa Creu i Sant pau, Barcelona
  - Hospital Juan Roamon Jimenez, Huelva
  - Hospital Universitario virgen de la arrixaca, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital virgen de la salud., Toledo
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Meixoiero, Vigo
- Switzerland (5):
  - Hôpital Fribourgeois, Fribourg
  - Centre hospitalier universitaire vaudois, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
- United Kingdom (6):
  - Brighton and Sussex Hospitals, Brighton
  - Craigavon Cardiac Center, Craigavon
  - Guy's and St.Thomas'Hospitals, London
  - King's College London, London
  - Freeman Hospital, Newcastle upon Tyne
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varenne O, Cook S, Sideris G, Kedev S, Cuisset T, Carrie D, Hovasse T, Garot P, El Mahmoud R, Spaulding C, Helft G, Diaz Fernandez JF, Brugaletta S, Pinar-Bermudez E, Mauri Ferre J, Commeau P, Teiger E, Bogaerts K, Sabate M, Morice MC, Sinnaeve PR; SENIOR investigators. Drug-eluting stents in elderly patients with coronary artery disease (SENIOR): a randomised single-blind trial. Lancet. 2018 Jan 6;391(10115):41-50. doi: 10.1016/S0140-6736(17)32713-7. Epub 2017 Nov 1. PMID 29102362